CLINICAL TRIAL: NCT01910805
Title: Lifestyle Intervention for African-American Women: A Pilot Study for Women With a Recent History of Gestational Diabetes (The LIFe Study)
Brief Title: Recent GDM Lifestyle Intervention
Acronym: LIFe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Tamarra James-Todd, Associate Epidemiologist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 108628
Record Dates: First submitted 2013-07-17; First posted 2013-07-30 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes Mellitus; Diabetes, Gestational
Keywords: Gestational diabetes; Diabetes mellitus; diabetes in pregnancy; diabetes risk; diabetes risk awareness; African-American; Women
MeSH Terms: conditions — Diabetes Mellitus; Diabetes, Gestational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle and Risk Awareness class (Experimental): Women will attend a 3- and 9-month postpartum group nutrition and physical activity education class.
  Interventions: Behavioral: Lifestyle and Risk Assessment class
- Standard Care (No Intervention): Women will receive standard postpartum care for gestational diabetes mellitus.

INTERVENTIONS:
Behavioral: Lifestyle and Risk Assessment class — Classes will be conducted by a CITI-certified Boston Public Health Commission nutritionist, who is a consultant on this project and has previously worked within the Boston African-American community to increase diabetes awareness and reduce diabetes risk. These classes will be held at a local community center to provide maximal accessibility to the women.
  The intervention group will attend classes mentioned at the aforementioned centers. Each class will take 2-hours and be conducted by a CITI-certified registered nutritionist with extensive knowledge of working in the African-American community. Both classes will include a cooking demonstration. In addition, the class will include a tour of a local supermarket to aid women in identifying healthy food choices.
  Arms: Lifestyle and Risk Awareness class

SUMMARY:
Women with a history of gestational diabetes (GDM) have a substantially increased risk of developing type 2 diabetes. In fact, 50-70% of these women will go on to develop type 2 diabetes within the 20 years following their GDM-complicated pregnancy. Perceived risk of developing type 2 diabetes among women with a history of GDM may be particularly important to altering behavior changes associated with reducing risk. Certain populations have lower perceived risk of developing type 2 diabetes, despite having a higher prevalence of the disease. Specifically, African-Americans have a lower perceived risk of developing type 2 diabetes compared to whites, despite their more than doubled risk of developing the disease. Improvement in awareness of diabetes risk among African-American women at high-risk of developing type 2 diabetes, such as those with a history of GDM, could reduce future risk of this disease among this group.

As such, we will conduct a two-armed, pilot randomized controlled trial to evaluate whether a postpartum diabetes education intervention, incorporating nutrition, exercise, and diabetes risk assessment can improve diabetes risk awareness, diet, and physical activity levels at 1-year post-pregnancy among African-American women with a recent history of gestational diabetes.

We hypothesize that attendance at a 3-month and 9-month postpartum diabetes education class will:

1. Improve diabetes awareness as measured using the Risk Perception for Developing Diabetes among women in the intervention group compared to women in the control group when measuring at 3-months postpartum compared to 12-months postpartum
2. Improve dietary habits and physical activity levels in the intervention group compared to the control group when measuring at 3-months postpartum compared to 12-months postpartum

DETAILED DESCRIPTION:
Study subjects will be recruited from the Brigham and Women's Hospital's (BWH)Diabetes and Pregnancy Program. Obstetricians will assist in the study by introducing the study to women with gestational diabetes (GDM), who are currently in their third trimester of pregnancy and asking the women to which race/ethnicity do they self-identify. Those women who self-identify as Black or African-American will be told by their health care provider that a Research Assistant from our study would like to speak with them about our study after their appointment and that the study is only for research purposes and is not mandatory for their treatment or care at BWH, but is on voluntary basis only.

Our Research Assistant will approach all women who self-identify as African-American and have GDM, who are in their third trimester (as identified by the obstetrician). For women who are interested in learning more about the study, but do not have time to hear more about it during the initial contact, the Research Assistant will obtain their contact information to describe the study and discuss the woman's possible participation at a later point in time.

For those women who have time to learn more about the study immediately following their obstetrics appointment at BWH, our Research Assistant will take women into a private room within the obstetrics clinic and provide them with general information about the study. If a woman is interested, we will ask the woman a set of screening questions to assess their eligibility. The screening questions will not include any personal identifying information and will only be collected to determine eligibility and response rates. If eligible for participation in our study, we will collect the eligible woman's contact information and provide the woman with an informed consent form to be reviewed and signed either at that time to our Research Assistant or returned to us by mail using a provided stamped, addressed envelope within 2 weeks of having received the form. Description of the study, confirmation of contact information, administration of the screening questionnaire, and receipt and review of consent documents will occur similarly by phone for those women who were not available to learn more about the study immediately following their obstetrics visit, but who expressed interests in learning more about the study at a later time point.

Given that women have until 3 months post-pregnancy to be enrolled in our study, we will also use a flyer with a detachable card and a brochure to try to recruit women during their 6-week postnatal visit, as well as at the time of delivery, during their hospital stay. These additional recruitment time points will maximize recruitment efforts. Recruitment at the 6-week postnatal visit will be similar to that described above for the third trimester clinic visit. For those women that we attempt to recruit at the time of delivery, we will have an obstetrician notify us of a delivering woman, who has self-identified as African-American and had GDM during her recent pregnancy. Our Research Assistant will approach women on the Labor and Delivery floor after the woman's delivery. At this time the study will be explained to her and the woman will be asked to answer screening questions, if she is interested in the study. An informed consent will be provided, if the woman is eligible. The woman can either complete the informed consent at that time or return it to our study staff within 2 weeks.

Upon return of the signed informed consent form, we will enroll the woman in the study and randomize her to receive either the study intervention or standard care. We will ensure balance in this process through the use of block randomization. At this time point, our research assistant will assist with scheduling the woman's 6-week postpartum follow-up visit, which is a part of her standard medical care. This assistance with scheduling, will aid in making sure that the potential study participant receives her 6-week postpartum diabetes screening. If she fails the screening, then she will be notified by a study clinician and withdrawn from the study.

For women who do not return the consent form within 2-weeks of having initially received it from our research assistant, we will re-contact the woman to follow-up with her about her interest in participating in the study. Eligible women will be re-contacted either by phone or e-mail, based on the woman's preferred method of contact, up to three times, to obtain the informed consent. After the third unsuccessful re-contact, we will stop attempts to obtain the consent form. We will also not re-contact a woman, if they state they are no longer interested in the study.

Again, as a part of enrollment into the study, we will obtain e-mail addresses and mailing addresses of our study participants (see Script C1). We will also obtain telephone information in order to call or text the woman, if this is her preferred contact method. At 3-months we will send a secure web link for completion of the 3-months web-based questionnaire to be completed by the woman. For women without internet access or those who do not wish to complete the questionnaire online, we will mail a paper-version of the questionnaire at 3-months postpartum. Likewise, a web link or paper questionnaires will be sent at 6-months, 9-months, and 12-months postpartum. If we have not received the completed questionnaire, we will contact the study participant by phone to determine whether she received the initial questionnaire and if she has any questions. All women enrolled in the study (both the intervention group and standard care group) will be asked to complete these questionnaires. We will also send a text reminder for those women who listed text as a preferred method of contact.

For those women enrolled in the intervention arm, the research assistant will contact them via phone to schedule them for their 3-month and 9-month class to be held at a local community centers. Two weeks before the class we will send a reminder card either via e-mail, text message, or postal mail. Two days before the class our Research Assistant will contact the women by phone to remind them of the class, location, and time. Women will also be reminded at this time to bring a favorite recipe to the class.

The intervention group will attend classes mentioned at the aforementioned centers. Each class will take 2-hours and be conducted by a Collaborative Institutional Training Initiative (CITI) certified registered nutritionist familiar with working in the GDM population and with extensive experience working in the African-American community. Both classes will include a cooking demonstration. In addition, the class will include a tour of a local supermarket to aid women in identifying healthy food choices. The classes will cover the following material:

3-month class:

1. Introductions: Nutritionist/Life coach will introduce herself and will encourage others to introduce themselves on a first name basis only.
2. Overview of class and class guidelines: Nutritionist/Life coach will provide an overview of the material to be covered as well as class guidelines
3. Diabetes Risk Awareness: Focus on diabetes risk factors, as well as symptoms of diabetes, and lifestyle factors that can reduce diabetes risk.
4. Review Weight Loss Goals: Subjects will weigh in at each visit: Discuss the benefit of weight loss on the reduction of risk of future type 2 diabetes in the mom.
5. Good Nutrition, Healthy Plate and Portions: Review portion sizes using handouts. There will also be a focus on adding fruits and vegetables, learning about healthy versus unhealthy fat, as well as label reading.
6. Infant feeding: Review/discuss the benefits of breastfeeding for mom and the baby including reducing maternal weight retention, and reducing infant and child obesity. Review optimal timing of introduction of solid foods and types of foods healthy for your child.
7. Ways to reduce your diabetes risk: Discussion of lifestyle factors that can reduce your diabetes risk, including physical activity and sleep.
8. Exercise Basics: Review options for moderate intensity cardiovascular exercise and strength training, including walking and the use of resistance bands, and discuss exercise goals.
9. Making Your Recipes Healthy: Focus on adapting popular recipes, as well as those of study participants to make them healthy. Participants will be asked to submit one favorite family recipe at the beginning of the study. The group will work together to modify all the recipes using healthy substitutions.
10. Cooking Demonstration: The nutritionist/group teacher will prepare a healthy meal during the class time. This will showcase healthy food choices, measuring and food preparation skills, as well as methods of cooking. Class participants will be welcomed to partake in the meal, once prepared.

9 month class:

1. Review of Diabetes and Diabetes Risk Awareness: Review diabetes risk factors, prevention measures used to reduce diabetes risk, and signs and symptoms of diabetes.
2. Review Weight Loss Goals: Subjects will weigh in at this time point and discuss the benefits of weight loss on the reduction of risk of future type 2 diabetes in the mom.
3. Eating Healthy, Healthy Plate and Portions: Review portion sizes using handouts. We will re-emphasize the importance of adding fruits and vegetables, and discuss healthy and unhealthy fats based on current dietary habits. Also, focus on label reading
4. Supermarket Smarts, Label reading and Dining Out: Tips for making healthy choices at the grocery store. Review how to make healthier choices when dining out, with instruction including a sample restaurant menu. In addition, participants will become familiar with how to read food labels.
5. Assessment of barriers to healthy lifestyle: Participants will discuss with nutritionist/group teacher issues surrounding healthy eating, barriers to physical activity and other healthy lifestyle behaviors associated with reduced risk of diabetes. Discussion will focus on solutions to overcoming these barriers.
6. Cooking Demonstration: The nutritionist/group teacher will provide a prepare and cook a health meal during the class time. This will showcase healthy food choices, measuring and food preparation skills, as well as methods of cooking. Class participants will be welcomed to partake in the meal, once prepared.

For women in the intervention group, onsite childcare at the Boys and Girls Club will be made a possible option through the use of already-certified childcare providers. We will also offer women the option of covering childcare at home for 4-hours (to cover commuting time, as well as the time for the 2-hour class) per session. Description of this compensation will be discussed below. If necessary, women will be allowed to bring their infant children to the class to ensure the woman is able to attend.

Upon completion of the class, the woman will be asked a set of qualitative questions regarding the class information and structure to better inform a larger, future intervention.

ELIGIBILITY:
Inclusion Criteria:

* Have gestational diabetes during current or most recent pregnancy
* Be less than 3 months postpartum
* Age between >=18 years
* Preconception BMI <45
* Singleton pregnancy
* Self-identified Black/African-American race/ethnicity
* Speak English

Exclusion Criteria:

* Preexisting diabetes or diabetes diagnosed at the 6 week 75 gram oral glucose tolerance test.
* BMI >=45.
* Multiple gestation (i.e. twins, triplets, etc.)

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in Diabetes Risk Awareness from baseline to 12 months postpartum | 3-12 months postpartum
  Using an adapted version of the Risk Perception Survey for Developing Diabetes for women with a history of gestational diabetes, women will be asked to respond on web-based or paper questionnaires regarding their individual and group risk of getting diabetes. The primary outcome will measure the change in their awareness of diabetes based on their diabetes risk perception score at baseline (3 months postpartum) compared to 12 months postpartum.

SECONDARY OUTCOMES:
Change in diet patterns from baseline to 12 months postpartum | 3 months to 12 months postpartum
  Women will be asked to respond to a adapted food frequency questionnaire. This food frequency questionnaire has been previously used in postpartum populations and is correlated with various health outcomes in observational studies. Diet information will be asked using the same food frequency questionnaire multiple times and the difference between baseline (3 months postpartum) and 12 months postpartum will be measured.
Change in physical activity levels from baseline to 12 months postpartum | 3 to 12 months postpartum
  Women will be asked to respond to questions regarding their physical activity level using an adapted physical activity questionnaire from the Nurses' Health Study. These questions will be adapted for use in a postpartum, African-American population. Women will be asked about their physical activity levels multiple times and the difference between physical activity levels at baseline (3 months) and at 12 months postpartum will be measured.

OTHER OUTCOMES:
Change in diabetes risk awareness from baseline to 9 months | 3 months to 9 months postpartum
Change in diet patterns from baseline to 9 months postpartum | 3 months to 9 months postpartum
Change in physical activity levels from baseline to 9 months postpartum | 3 months to 9 months postpartum
Change in diabetes risk awareness from baseline to 6 months postpartum | 3 to 6 months postpartum
Change in diet patterns from baseline to 6 months postpartum | 3 to 6 months postpartum
Change in physical activity levels from baseline to 6 months postpartum | 3 to 6 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Tamarra James-Todd, PhD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States